CLINICAL TRIAL: NCT06100497
Title: Efficacy and Safety of PD-1 Inhibitor Combined With Chemotherapy in Locally Advanced (III-IVB) Poorly Differentiated Head and Neck Squamous Cell Carcinoma: a Multi Cohort, Prospective Phase II Study
Brief Title: Efficacy and Safety of PD-1 Plus Chemotherapy in Poorly Differentiated Locally Advanced (LA) HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-001
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage IVB cohort (Experimental): patients must undergo evaluation after receiving 2 cycles of PD-1 (pembrolizumab, 200mg, IV, Q3W) combined with platinum-based (cisplatin: 75 mg/m2, IV, Q3W) and albumin paclitaxel (260mg/m2, IV, Q3W) treatment (Arm 1 may receive a third cycle of treatment based on tumor regression). if achieving CR/PR on imaging, suitable for surgical treatment, not suitable for surgery or SD/PD patients, subsequent synchronous chemoradiotherapy or synchronous chemoradiotherapy combined with PD-1 (pembrolizumab) treatment (total of no more than 17 cycles).
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Paclitaxel-albumin
- Stage III-IVA cohort (Experimental): patients with stage III and IVA (T3NxM0, T4aNxM0) receive PD-1 (pembrolizumab, 200mg, IV, Q3W) combined with platinum-based chemotherapy (cisplatin: 75 mg/m2, IV, Q3W) and albumin-bound paclitaxel (260mg/m2, IV, Q3W) for 2 cycles. Patients who undergo surgery within 2 weeks based on pathological results are given PD-1 monotherapy maintenance treatment or low-dose radiotherapy followed by PD-1 monotherapy maintenance treatment if they achieve pathological complete response (pCR). Non-pCR patients with positive surgical margins or extracapsular extension after surgery receive PD-1 maintenance treatment after concurrent chemoradiotherapy (up to a maximum of 17 cycles). Patients without high-risk factors receive PD-1 maintenance treatment after radiotherapy (up to a maximum of 17 cycles).
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Paclitaxel-albumin

INTERVENTIONS:
Drug: Pembrolizumab — Mainly used for neoadjuvant treatment and subsequent adjuvant or maintenance treatment
Drug: Cisplatin — Mainly used for neoadjuvant treatment and concurrent chemoradiotherapy
Drug: Paclitaxel-albumin — Mainly used for neoadjuvant treatment
  Other Names: albumin paclitaxel

SUMMARY:
Patients with locally advanced (stage III to stage IVB) poorly differentiated head and neck squamous cell carcinoma (excluding nasopharyngeal carcinoma) who meet the inclusion criteria will have their blood samples collected, tumor tissue samples or patient paraffin tissue, and slides for comprehensive genomic sequencing and analysis. The study is divided into two groups. Arm1 group: Patients with stage IVB (T4bNxM0) poorly differentiated head and neck squamous cell carcinoma (excluding nasopharyngeal carcinoma) will receive PD-1 combined with platinum-based chemotherapy and albumin-bound paclitaxel (dose according to the drug instructions) for 2 to 3 cycles (determined by the researcher based on tumor shrinkage). If the imaging achieves complete response (CR) or partial response (PR), suitable patients will undergo surgical treatment. Patients who are not suitable for surgery or have stable disease (SD)/progressive disease (PD) will receive concurrent chemoradiotherapy or concurrent chemoradiotherapy combined with PD-1 treatment (up to a total of 17 cycles). Arm2 group: Patients with stage III and IVA (T3NxM0, T4aNxM0) poorly differentiated head and neck squamous cell carcinoma (excluding nasopharyngeal carcinoma) will receive PD-1 combined with platinum-based chemotherapy and albumin-bound paclitaxel (dose according to the drug instructions) for 2 cycles. Patients who undergo surgery within 2 weeks will receive PD-1 monotherapy maintenance treatment or low-dose radiotherapy followed by PD-1 monotherapy maintenance treatment based on pathological results. Patients who do not achieve pathological complete response (pCR) and have positive surgical margins or extracapsular extension will receive concurrent chemoradiotherapy followed by PD-1 maintenance treatment (up to a total of 17 cycles). Patients without high-risk factors will receive PD-1 maintenance treatment after radiotherapy (up to a total of 17 cycles). After completion of treatment, all patients will be followed up every 3 months for 1 year. Subsequently, patients will be followed up every 6 months for 3 years. Thereafter, patients will be followed up annually. Patient recurrence and survival data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced (III-IVB) poorly differentiated head and neck tumors (hypopharyngeal cancer, laryngeal cancer, oropharyngeal cancer, nasal cavity and sinus cancer, excluding nasopharyngeal cancer) with a confirmed diagnosis by histology and/or cytology;
* Patients who can receive systemic treatment or PD-1/L1 monotherapy before treatment;
* Patients in arm2 must be evaluated as having resectable tumors before treatment;
* The investigator believes that the patient can safely receive PD-1 combined with platinum-based and albumin-bound paclitaxel treatment;
* Age ≥ 18 years;
* ECOG (Eastern Cooperative Oncology Group) 0-1；
* Measurable disease defined by RECIST v1.1;
* Adequate bone marrow reserve and organ function: absolute neutrophil count (ANC) ≥ 1,000/μL, platelets ≥ 75,000/μL, hemoglobin ≥ 8g/dL, no transfusion or erythropoietin (EPO) dependence (within 7 days of assessment);
* Renal function: serum creatinine ≤ 1.5X upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 60mL/min, creatinine level > 1.5X institutional ULN. (GFR can also be used instead of creatinine or CrCl). Creatinine clearance should be calculated according to institutional standards;
* Liver function: For subjects with total bilirubin levels >1.5 ULN, serum total bilirubin ≤1.5X ULN or direct bilirubin ≤ULN; For patients with liver metastasis, aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5X ULN or ≤5X ULN; Albumin > 2.5 mg/dL;
* Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5X ULN, if subjects require anticoagulant therapy, PT or PTT (partial thromboplastin time) should be within the allowable range of anticoagulant use;
* Women should agree to use contraception during the study and for 6 months after the end of the study (such as intrauterine devices (IUDs), contraceptive pills, or condoms); Within 7 days before study enrollment, serum or urine pregnancy test should be negative, and patients must be non-lactating; Men should agree to use contraception during the study and for 6 months after the end of the study.

Exclusion Criteria:

* Patients who have previously received PD-1/L1 combined chemotherapy drugs;
* Patients with a history of other malignant tumors (including unknown primary) within the past 5 years. Note: Excluding stage 1 or 2 skin basal/squamous cell carcinoma or in situ carcinoma receiving potentially curative treatment;
* Patients who cannot tolerate postoperative radiotherapy;
* Patients known to be allergic to the study drug or its active ingredients or excipients;
* Patients with any unstable systemic diseases, including but not limited to: severe infection, uncontrolled diabetes, unstable angina, cerebrovascular accident or transient ischemic attack, myocardial infarction, congestive heart failure, severe -Patients with underlying immune deficiencies, chronic infections, including HIV, hepatitis, tuberculosis (TB), or autoimmune diseases;
* Patients with potential hematologic issues, including bleeding diathesis, known prior gastrointestinal bleeding requiring intervention within the past 6 months, active pulmonary embolism or deep vein thrombosis (DVT) unstable on anticoagulation regimen;
* History or evidence of active non-infectious pneumonia;
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Subjects with prior treated brain metastases may participate as long as they are stable (no evidence of imaging progression for at least four weeks prior to the first trial treatment and any neurological symptoms have returned to baseline), no new or enlarging brain metastases, and no use of steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which will be excluded regardless of clinical stability;
* Within 7 days before the first day of the first cycle, at the same time (or receiving) treatment with drugs that may affect drug metabolism;
* Pregnant or breastfeeding, or expecting to become pregnant or give birth during the expected trial period;
* Any uncontrolled concurrent disease, including but not limited to persistent or active infection, symptomatic congestive heart failure, unstable angina, arrhythmia;
* Screening EKG> 475 ms prolonged corrected QT (QTc) interval;
* Ejection fraction <40% by 2D echocardiogram (ECHO) during screening;
* Any serious medical or mental illness/symptoms, including substance use disorders, may interfere with or limit compliance with study requirements/treatments in the investigator's judgment;
* Having active autoimmune diseases requiring systemic treatment in the past 2 years (even with disease-modifying agents, corticosteroids, or immunosuppressive drugs). Alternative therapies (e.g., thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered a form of systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 month
  The proportion of subjects with best overall response (BOR) assessed as complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  Defined as the time from randomization to the date of first disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | 6 month
  According to RECIST v1.1 criteria, it assesses the proportion of subjects with complete response (CR), partial response (PR), and stable disease (SD) in terms of overall best response (BOR).
Time to objective response (TTR) | 3 years
  Defined as the duration from the start of medication to the date of first documented CR or PR (whichever occurs first). Tumor response is based on confirmed tumor response, and the response date is from the first observation, not the confirmed response.
Duration of Response (DOR) | 3 year
  The duration from the date of first assessment as CR or PR to the date of first assessment as disease progression or death for subjects who achieved complete response or partial response (CR or PR).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT06100497/Prot_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT06100497/ICF_001.pdf